CLINICAL TRIAL: NCT03547284
Title: The Role of Sugarless Gum Chewing in Regaining Bowel Motility in Patients Undergoing Cesarean Section
Brief Title: the Role of Gum Chewing in Regaining Bowel Motility in Patients Undergoing Cesarean Section
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona M Shaban, associate obgyn professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Woman Health University Egypt
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Effect of Gum Chewing on Regaining Bowel Motility After Cesarean Section

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 81 patients,group 1 (Active Comparator): 81 women will receive 1 stick of sugarless gum for 15 minutes every 2 hours after surgery .
  Interventions: Drug: sugarless gum
- 81 patients,group 2 (No Intervention): 81 patients will have traditional management(oral intake of clear fluids after hearing of first intestinal sounds or passage of flatus and regular diet after passage of stool)

INTERVENTIONS:
Drug: sugarless gum — 81 patients will receive 1 stick of sugarless gum(Samara gum) for 15 minutes every 2 hours
  Other Names: Samara Gum
  Arms: 81 patients,group 1

SUMMARY:
Aim:to evaluate the efficacy of postoperative gum chewing on the recovery of bowel motility after cesarean section.

DETAILED DESCRIPTION:
this study will be conducted on 162 patients undergoing cesarean section in obstetrics and gynecology department at Kasr el Ainy Hospital,Kairo university.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35

  --Spinal anesthesia
* Pfannensteil incision

Exclusion Criteria:

* History of drug consumption especially opioids
* water and electrolyte disturbance
* History of abdominal surgery except cesarean section
* Intra and severe post operative complications
* diabetes
* Pre-eclampsia
* Hypothyroidism
* Muscular and neurological disorder
* Inability to chew gums

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
first bowel sound in hours | 4-6 hours

SECONDARY OUTCOMES:
first passage of flatus in hours,the first defecation in hours | 4-6 hours

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo University Hospital,obstetrics and gynecology departement, Egypt, Cairo
  - Woman's Health University Hospital, Egypt, Cairo